CLINICAL TRIAL: NCT00119444
Title: Evaluation of Acetabular Perfusion After Ganz Osteotomy by Positron Emission Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050606
Record Dates: First submitted 2005-07-05; First posted 2005-07-13 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2009-09

CONDITIONS: Osteoarthritis
Keywords: PET; Periacetabular osteotomy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- periacetabular osteotomy (Other)
  Interventions: Procedure: Periacetabular osteotomy

INTERVENTIONS:
Procedure: Periacetabular osteotomy — osteotomy of the pelvis to increase acetabular coverage
  Other Names: PAO

SUMMARY:
The purpose of this study is to examine the blood flow in acetabulum after periacetabular osteotomy by Positron Emission Tomography (PET).

DETAILED DESCRIPTION:
As a consequence of periacetabular osteotomy the blood flow in acetabulum is decreased. After periacetabular osteotomy has been performed there is fine contact between the osteotomised acetabulum and the rest of the pelvis and the potential for healing is good. However, it has not been investigated how much the blood flow in acetabulum is changed after surgery. The blood flow is considered to be vital for how the pelvis heals after surgery. Most likely, the blood flow is important in relation to which degree osteoarthritis can be prevented after periacetabular osteotomy.

It is possible to estimate the blood flow by Positron Emission Tomography of the dysplastic hip joint pre- and postoperatively. In this study the blood flow and fluoride uptake is quantified by Positron emission tomography based on measurements of O-15 water and F-18 fluoride.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiologically diagnosed hip dysplasia (CE-angle < 25°).
* Patients with osteoarthritis graded 0, 1 or 2 defined according to Tönnis' classification. Patients with pain from hip
* Age > 18 years.
* Minimum 110° flexion in hip joint and closed growth zones in the pelvic.
* Informed consent.

Exclusion Criteria:

* Patients with neurological diseases
* Patients with calvé-Legg-Perthes syndrome.
* Patients where an femoral intertrochanteric osteotomy is necessary.
* Patients with medical sequelae after earlier hip surgery.
* Females who are pregnant.
* Patients with metal implants.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2004-01; Primary Completion 2008-01 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
changes in blood flow | within the first three weeks after operation

SECONDARY OUTCOMES:
fluoride uptake | within the first three weeks after operation

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, MD, Prof., Principal Investigator — Orthopaedic Center, Aarhus University Hospital, Aarhus, Denmark
Locations (1):
- Orthopaedic Center, Aarhus University Hospital, Aarhus, Denmark